CLINICAL TRIAL: NCT01878760
Title: APRICOT: Anaesthesia PRactice In Children Observational Trial - European Prospective Multicenter Observational Study: Epidemiology of Severe Critical Events in Paediatric Anaesthesia
Brief Title: APRICOT: Anaesthesia PRactice In Children Observational Trial
Acronym: APRICOT
Status: Completed | Type: Observational
Sponsor: European Society of Anaesthesiology (Other)
Responsible Party: Sponsor
Other Study IDs: APRICOT
Record Dates: First submitted 2013-05-28; First posted 2013-06-17 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Anaesthesia; Children
Keywords: APRICOT; Anaesthesia; Children; kids; Paediatric Anaesthesia; Observational Trial; epidemiology; severe critical events in; European Society of Anaesthesiology; Europe

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aims of the APRICOT study are:

* To establish the incidence of severe critical events in children undergoing anesthesia in Europe.
* To describe the differences in paediatric anaesthesia practice throughout Europe.
* To study the potential impact of this variability on the occurrence of severe critical events (Laryngospasm, Bronchospasm, Pulmonary aspiration, Drug error, Anaphylaxis, Cardiovascular instability, Neurological damage, Perianaesthetic cardiac arrest and postanaesthetic Stridor).

DETAILED DESCRIPTION:
Despite the introduction of better-structured programmes for paediatric anaesthesia training and the development of some recommendations for paediatric anaesthesia services, the incidence of severe critical events in children is still unknown in Europe. Considering that the major life-threatening complications following general or regional anaesthesia are uncommon, it is therefore crucial to consider a large multinational, multicentre trial in order to establish a realistic statistical estimation and identify the risk factors for severe critical events. Thus, this prospective observational multicentre cohort study is designed to identify the incidence and potential risk factors of severe critical events in children undergoing anaesthesia in Europe.

The study aims to include all children from birth to 15 years old scheduled for an elective or urgent diagnostic or surgical procedure under sedation or general anaesthesia with or without regional analgesia or under regional anaesthesia. This represents the denominator dataset for calculation of the incidence of severe critical events, which is the primary aim of the study. The anaesthesiologist in charge will record the occurrence of selected severe critical events during and up to 60 minutes after anaesthesia or sedation AND requiring immediate intervention. These severe critical incidents include: Laryngospasm, Bronchospasm, Pulmonary aspiration, Drug error, Anaphylaxis, Cardiovascular instability, Neurological damage, Perianaesthetic cardiac arrest and postanaesthetic Stridor. The secondary endpoint is represented by the risk factors and the consequences for the occurrence of these severe critical events including in-hospital mortality established up to 30 days or at discharge. Relevant aspects of the child's medical and family history will be recorded.

Following sample size estimation, we plan to recruit at least 25 000 children over a period of two consecutive weeks including weekends and after-hours across the 30 European countries represented at the European Society of Anaesthesiology Council or part of geographical Europe. The 2-week recruitment period will be chosen by each site commencing on 15 March 2014.The last possible inclusion date will be decided by the Study Steering Committee depending on the recruitment rate. Participating hospitals will be provided with data acquisition sheets that enable anonymous standardized recording of all patients' parameters, which will be used by the local institution to fill in the electronic case report form (eCRF).

Descriptive statistical analysis will be performed for the primary endpoint (occurrence of severe critical events and 95% confidence interval). Univariate and multivariate analysis will be performed to test factors associated with the endpoint. Results of logistic regression will be reported as adjusted odds ratio (OR) with 95 % confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* Age: from birth to 15 years included
* All children admitted for an inpatient or outpatient procedure under general anaesthesia with or without regional analgesia or under regional anaesthesia alone. This includes all kind of surgeries and procedures requiring anaesthesia and analgesia to be performed such as central venous access, burn care, cast, etc.,
* Children admitted for a diagnostic procedure under sedation (performed by an Anaesthetist) or general anaesthesia (such as endoscopy, radiology (CT-scan, MRI), cardiac catheterisation and electrophysiology, PET-scan, radiotherapy, lumbar and bone marrow puncture, biopsies), diagnostic procedure under general anaesthesia (such as endoscopy, radiology…)
* Children admitted for urgent or emergency procedure performed in- or out-of-hours.

Exclusion Criteria:

* Children admitted directly from the intensive care units to the operating rooms
* Anaesthesia procedures in the neonatal or paediatric intensive care units.
* Age: All children aged ≥ 16 years.

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children from birth to 15 years included admitted for an inpatient or outpatient procedure under general anaesthesia with or without regional analgesia or admitted for a diagnostic procedure under general anaesthesia (such as endoscopy, radiology…) or admitted out-of-hours for emergency procedures
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Incidence of severe critical events | Children will be followed for the duration of their anaesthesia procedure and up to 60 minutes afterwards
  Incidence of the following severe critical events defined as any incident occurring during and up to 60 minutes after anaesthesia or sedation (PACU), requiring immediate intervention and that may lead to major disability and/or death:
  * Laryngospasm
  * Bronchospasm
  * Pulmonary aspiration
  * Drug error
  * Anaphylaxis
  * Cardiovascular instability
  * Neurological damage
  * Perianaesthetic Cardiac arrest
  * Postanaesthetic Stridor (in the PACU)

SECONDARY OUTCOMES:
Risk factors for the occurrence of severe critical events | Children will be followed for the duration of their anaesthesia procedure and up to 60 minutes afterwards
  Assessment of risk factors will be achieved by collecting data on social and demographic data of the patients, family and child's medical history, presence of co-morbidities, details on anesthesia procedure, elective or emergency cases, level of experience of the anesthesiologist, postoperative prescriptions.
Consequences of the critical events: irreversible damage, in-hospital mortality | in-hospital and up to 30 days
  Consequences of critical events: no harm, minor sequelae, irreversible damage, in-hospital mortality (up to 30 days or discharge).

CONTACTS AND LOCATIONS:
Overall Officials: Walid Habre, M.D., Study Chair — University Hospital, Geneva; Francis Veyckemans, M.D., Study Director — Cliniques Universitaires St Luc asbl Brussels
Locations (38):
- Medical University Graz, Graz, Austria
- Cliniques Universitaires St Luc, Brussels, Belgium
- General Hospital Pula, Pula, Croatia
- University Children´s Hospital, Brno, Czechia
- Odense University Hospital, Odense, Denmark
- Tartu University Hospital, Tartu, Estonia
- Finland (2):
  - Oulu University Hospital, Oulu
  - Turku University Hospital, Turku
- France (2):
  - CHU Lille, Lille
  - Lapeyronie University Hospital, Montpellier
- Germany (3):
  - Universitaetsklinikum Leipzig, Leipzig
  - Cnopf'sche Kinderklinik/Klinik Hallerwiese, Nuremberg
  - Asklepios Klinik Sankt Augustin GmbH - Department of Paediatric Anaesthesia, Sankt Augustin
- Gibraltar Health Authority, St. Bernard´s Hospital, Gibraltar, Gibraltar
- Children Hospital P&A Kyriakoy, Athens, Greece
- Our Ladys Children's Hospital, Dublin, Ireland
- Schneider Children's Medical center of Israel, Petah Tikva, Israel
- Instituto Giannina Gaslini, Genoa, Italy
- University Clinical Center of Kosovo, Pristina, Kosovo
- Children University Hospital, Riga, Latvia
- Vilnius Children Hospital, Vilnius, Lithuania
- Mater Dei Hospital MSD, Msida, Malta
- Maastricht University Medical Center MUMC, Maastricht, Netherlands
- Oslo University Hospital, Rikshospitalet, Oslo, Norway
- Clinical University Hospital Department of Anaesthesiology and Intensive Care, Wroclaw, Poland
- Centro Hospitalar Lisboa Norte - Hospital de Santa Maria, Lisbon, Portugal
- Spitalul de Copiin Maria Curie, Bucharest, Romania
- Pirogov Russian National Research Medical University, Moscow, Russia
- University Childrens hospital, Belgrade, Serbia
- Paediatric District Hospital, Banská Bystrica, Slovakia
- University Klinical Centre Ljubljana, Ljubljana, Slovenia
- Hospital Sant Joan Déu, Esplugues de Llobregat, Spain
- Queen Silvis Childrens Hospital Sahlgrens University Hospital, Gothenburg, Sweden
- Switzerland (2):
  - Geneva University Hospitals, Geneva
  - Anästhesie Kinderspital Klinik für Anästhesie, Intensivmedizin, Rettungsmedizin und Schmerztherapie (KLIFAIRS) Luzerner Kantonsspital Spitalstrasse, Lucerne
- Cukurova University Faculty Of Medicine, Adana, Turkey (Türkiye)
- P.L.Shupyk National Medical Academy of Postgraduate Education, Municipal Children's Hospital #1, Kyiv, Ukraine
- Royal Hospital For Sick Children, Glasgow, Scotland, United Kingdom

REFERENCES:
- [Derived] Dagher K, Benvenuti C, Virag K, Habre W. The Incidence of Postoperative Complications Following Lumbar and Bone Marrow Punctures in Pediatric Anesthesia: Insights From APRICOT. J Pediatr Hematol Oncol. 2024 Apr 1;46(3):165-171. doi: 10.1097/MPH.0000000000002849. Epub 2024 Mar 4. PMID 38447107
- [Derived] Dahmani S, Laffargue A, Dadure C, Veyckemans F; French APRICOT trial group. Description of practices and complications in the French centres that participated to APRICOT: A secondary analysis. Anaesth Crit Care Pain Med. 2019 Dec;38(6):637-645. doi: 10.1016/j.accpm.2019.06.001. Epub 2019 Jun 11. PMID 31200009
- [Derived] Virag K, Sabourdin N, Thomas M, Veyckemans F, Habre W; APRICOT Group of the European Society of Anaesthesiology Clinical Trial Network. Epidemiology and incidence of severe respiratory critical events in ear, nose and throat surgery in children in Europe: A prospective multicentre observational study. Eur J Anaesthesiol. 2019 Mar;36(3):185-193. doi: 10.1097/EJA.0000000000000951. PMID 30640246
- [Derived] Engelhardt T, Virag K, Veyckemans F, Habre W; APRICOT Group of the European Society of Anaesthesiology Clinical Trial Network. Airway management in paediatric anaesthesia in Europe-insights from APRICOT (Anaesthesia Practice In Children Observational Trial): a prospective multicentre observational study in 261 hospitals in Europe. Br J Anaesth. 2018 Jul;121(1):66-75. doi: 10.1016/j.bja.2018.04.013. Epub 2018 May 18. PMID 29935596
- [Derived] Habre W, Disma N, Virag K, Becke K, Hansen TG, Johr M, Leva B, Morton NS, Vermeulen PM, Zielinska M, Boda K, Veyckemans F; APRICOT Group of the European Society of Anaesthesiology Clinical Trial Network. Incidence of severe critical events in paediatric anaesthesia (APRICOT): a prospective multicentre observational study in 261 hospitals in Europe. Lancet Respir Med. 2017 May;5(5):412-425. doi: 10.1016/S2213-2600(17)30116-9. Epub 2017 Mar 28. PMID 28363725